CLINICAL TRIAL: NCT07032298
Title: Phase I Clinical Study on the Safety, Pharmacokinetics and Antitumor Activity of SSGJ-612 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of SSGJ-612 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-612-101
Record Dates: First submitted 2025-06-19; First posted 2025-06-23 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SSGJ-612 (Experimental): In dose escalation phase, participants will receive one of the five increasing dose levels of SSGJ-612 respectively, intravenously (IV). During or after dose escalation, any dose levels that does not exceed the MTD can be expanded.
  Interventions: Drug: SSGJ-612

INTERVENTIONS:
Drug: SSGJ-612 — Intravenous injection

SUMMARY:
This study is an open-label phase I study to evaluate the safety, pharmacokinetics, and antitumor activity of SSGJ-612 in patients with advanced malignant solid tumors expressing HER2.

DETAILED DESCRIPTION:
The clinical trial consists of two phases. In the dose escalation stage, the accelerated titration method combined with the traditional "3+3" design will be adopted, to evaluate the safety and dose-limiting toxicity (DLT), and to determine the maximum tolerated dose (MTD) or the maximum dose of administration (MAD). In the dose expansion phase, several safe and effective dose levels of SSGJ-612 will be expanded and further evaluated in larger groups of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study, be willing to follow and complete all trial procedures, and sign the informed consent form;
2. Aged ≥18 and ≤75 years old at the time of signing the ICF, regardless of gender;
3. Expected survival ≥3 months;
4. Performance status (PS) score of 0-1 according to the Eastern Cooperative Oncology Group (ECOG) scale;
5. Patients with pathologically or cytologically confirmed locally advanced or metastatic malignant tumors who have failed standard treatment, are intolerant to standard treatment, or have no standard treatment available, and cannot undergo complete surgical resection or receive radical concurrent/sequential chemoradiotherapy;
6. Tumor tissue with HER2 expression;
7. At least one measurable tumor lesion assessed as the target lesion according to RECIST v1.1 criteria, and the lesion is suitable for repeated and accurate measurement.

Exclusion Criteria:

1. Presence of brainstem, meninges, or spinal cord metastasis, or spinal cord compression;
2. Presence of active central nervous system (CNS) metastatic lesions;
3. Individuals with clinical symptoms or requiring repeated drainage (once a month or more frequently) of pleural effusion, pericardial effusion, or ascites;
4. Primary or secondary immunodeficiency, including positive human immunodeficiency virus (HIV) test;
5. Known active tuberculosis; known active syphilis infection;
6. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
7. Use of any live vaccine or attenuated live vaccine within 4 weeks before the first dose, or plan to receive any live vaccine or attenuated live vaccine during the study;
8. Known severe allergic history to any component of the investigational drug, or history of severe allergic reaction to antibodies;
9. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | Through study completion, an average of 1 year
  Adverse Events (AEs) refers to all adverse medical events that occur in patients after they receive the investigational drug and do not necessarily have a causal relationship with the investigational drug. AEs were evaluated according to CTCAE V5.0.
Incidence of DLT | 14 days
  Dose-Limiting Toxicity

SECONDARY OUTCOMES:
ORR assessed by investigators per RECIST v1.1 | Through study completion, an average of 1 year
  Objective Response Rate (ORR) is the proportion of patients with Complete Response (CR) or Partial Response (PR), assessed by investigators per RECIST v1.1.
DoR assessed by investigators per RECIST v1.1 | Through study completion, an average of 1 year
  Duration of Response (DoR) is the time between the first onset of CR or PR and the first onset of Disease Progression (PD) (assessed by investigators per RECIST v1.1) or death from any cause.
DCR assessed by investigators per RECIST v1.1 | Through study completion, an average of 1 year
  Disease Control Rate (DCR) is the proportion of patients with CR, PR, and Stable Disease (SD), assessed by investigators per RECIST v1.1.
TTR assessed by investigators per RECIST v1.1 | Through study completion, an average of 1 year
  Time to Response (TTR) is the time from the start of treatment until the date of first documented response (assessed by investigators per RECIST v1.1).
PFS | Through study completion, an average of 1 year
  Progression-Free Survival (PFS) is the time between first initiation of study treatment to PD (assessed by investigators per RECIST v1.1) or death due to any reason.
OS | Through study completion, an average of 1 year
  Overall Survival (OS) is defined as the time from the start of treatment with SSGJ-612 until death due to any cause.
Cmax of SSGJ-612 | Through study completion, an average of 1 year
  Peak concentration (Cmax), in single dose period and multiple dose periods.
Cmin of SSGJ-612 | Through study completion, an average of 1 year
  Trough concentration (Cmin), in multiple dose periods.
Tmax of SSGJ-612 | Through study completion, an average of 1 year
  Peak time (Tmax), in single dose period and multiple dose periods.
T1/2 of SSGJ-612 | Through study completion, an average of 1 year
  Elimination phase half-life (T1/2), in single dose period and multiple dose periods.
AUC0-last | Through study completion, an average of 1 year
  Area under plasma concentration-time curve from 0 to the last quantifiable time point (AUC0-t), in single dose period and multiple dose periods.
Incidence of ADA and Nab | Through study completion, an average of 1 year
  Number of patients with detectable Anti-drug Antibody (ADA) and Neutralizing Antibodies (NAb).
The correlation between HER2 expression and efficacy | Through study completion, an average of 1 year
  The correlation between expression level of HER2 in tumor tissues and anti-tumor activity.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No